CLINICAL TRIAL: NCT06449547
Title: Risk Factors Analysis of Anxiety and Depression in Patients With Herpes Zoster Neuralgia and Characteristics of Serum Biomarkers and Functional Brain Magnetic Resonance Changes
Brief Title: Risk Factors of Anxiety and Depression in Patients With Herpes Zoster Neuralgia
Status: Recruiting | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, Deputy director of anesthesiology, Huazhong University of Science and Technology
Other Study IDs: TJ-IRB202401075
Record Dates: First submitted 2024-05-19; First posted 2024-06-10 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Herpes Zoster
Keywords: Anxiety; Depression; Herpes Zoster; Neuralgia
MeSH Terms: conditions — Herpes Zoster; Anxiety Disorders; Depression; Neuralgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum is obtained to test for biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- patients with anxiety: Patients in this group suffered from herpes zoster neuralgia and had a score more than or equal to 8 for Hospital Anxiety and Depression Scale- Anxiety questionnaire.
  Interventions: Diagnostic Test: Hospital Anxiety and Depression Scale
- patients without anxiety: Patients in this group suffered from herpes zoster neuralgia and had a score less than 8 for Hospital Anxiety and Depression Scale- Anxiety questionnaire.
  Interventions: Diagnostic Test: Hospital Anxiety and Depression Scale
- patients with depression: Patients in this group suffered from herpes zoster neuralgia and had a score more than or equal to 8 for Hospital Anxiety and Depression Scale- Depression questionnaire.
  Interventions: Diagnostic Test: Hospital Anxiety and Depression Scale
- patients without depression: Patients in this group suffered from herpes zoster neuralgia and had a score less than 8 for Hospital Anxiety and Depression Scale- Depression questionnaire.
  Interventions: Diagnostic Test: Hospital Anxiety and Depression Scale

INTERVENTIONS:
Diagnostic Test: Hospital Anxiety and Depression Scale — Hospital Anxiety and Depression Scale questionnaire is used to test patients for anxiety and depression.

SUMMARY:
The goal of this observational study is to explore risk factors of anxiety and depression in patients with herpes zoster neuralgia, and the changes of certain serum biomarkers and functional brain magnetic resonance images of these patients.

DETAILED DESCRIPTION:
Patients with herpes zoster neuralgia will be recruited and take Hospital anxiety depression rating scale (Hospital anxiety and 'scale, HADS) evaluation. According to the HADS Scores, patients will be divided into depression group and no depression, or anxiety group and no anxiety group. The clinical data the of two groups will be collected and statistically analyzed to explore the risk factors of anxiety and depression, including the changes of serum biomarkers and functional brain magnetic resonance imaging in patients with herpes zoster neuralgia accompanying anxiety or depression.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 18 years old
2. Diagnosed as herpes zoster neuralgia
3. Signing informed consent

Exclusion Criteria:

1. Unable to complete the scale assessment
2. History of mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in patients who are diagnosed as herpes zoster neuralgia
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
HADS score | during hospital stay, average of 1 week
  Enrolled patients will be first evaluated by Hospital Anxiety and Depression Scare questionaire and according to the HADS score, patients will be divided to group with anxiety/depression and group without anxiety/depression.

SECONDARY OUTCOMES:
Interleukin (IL）-1β plasma level | during hospital stay, average of 1 week
  Blood sample will be obtained from enrolled patients and the plasma level of inflammatory cytokines IL-1β （pg/ml）will be tested.
IL-2 receptor plasma level | during hospital stay, average of 1 week
  Blood sample will be obtained from enrolled patients and the plasma level of inflammatory cytokines IL-2 （u/ml）will be tested.
IL-6 plasma level | during hospital stay, average of 1 week
  Blood sample will be obtained from enrolled patients and the plasma level of inflammatory cytokines IL-6 （pg/ml）will be tested.
IL-8 plasma level | during hospital stay, average of 1 week
  Blood sample will be obtained from enrolled patients and the plasma level of inflammatory cytokines IL-8 （pg/ml）will be tested.
IL-10 plasma level | during hospital stay, average of 1 week
  Blood sample will be obtained from enrolled patients and the plasma level of inflammatory cytokines IL-10 （pg/ml）will be tested.
Interferon(INF)-α plasma level | during hospital stay, average of 1 week
  Blood sample will be obtained from enrolled patients and the plasma level of inflammatory cytokines INF-α （pg/ml）will be tested.
Brain-derived neurotrophic factor (BDNF) plasma level | during hospital stay, average of 1 week
  Blood sample will be obtained from enrolled patients and the plasma level of BDNF（pg/ml）will be tested.
C-reactive protein (CRP) plasma level | during hospital stay, average of 1 week
  Blood sample will be obtained from enrolled patients and the plasma level of CRP（mg/ml）will be tested.
Area under curve (AUC) of topological metrics of functional brain magnetic resonance imaging | during hospital stay, average of 1 week
  Functional brain magnetic resonance imaging will be performed in patients with anxiety or depression, and area under curve (AUC) of topological metrics including Eglob,Eloc,Cp,Lp,γ,λ and σ will be calculated and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Shuguang, M.D, Principal Investigator — Tongji medical college of Huazhong University of Science and technology
Locations (1):
- Tongji hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
no plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Background] Du J, Sun G, Ma H, Xiang P, Guo Y, Deng Y, Li S, Li X. Prevalence and Risk Factors of Anxiety and Depression in Patients with Postherpetic Neuralgia: A Retrospective Study. Dermatology. 2021;237(6):891-895. doi: 10.1159/000512190. Epub 2020 Dec 16. PMID 33326962